CLINICAL TRIAL: NCT04809090
Title: CO-ADAPT: Adaptive Environments and Conversational Agent Based Approaches for Healthy Ageing and Work Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tommaso Ciulli (Industry)
Collaborators: Università degli Studi di Trento (Other)
Responsible Party: Sponsor-Investigator, Tommaso Ciulli, Chief Research Officer, Idego srl
Organization: Idego srl (Industry)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: COADAPT 2019-2021
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Work Related Stress; Psychologic Adaptation
Keywords: work related stress; Psychological Adaptation
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: Subjects who will participate in the study voluntarily will be given some pre-intervention tests (T1) to assess their psychological well-being, to understand the main coping strategies they employ to manage stress, general stress, and the presence of cognitive impairment. Questionnaires will be used to collect data and exclude those subjects who do not meet the inclusion criteria.
  Subjects included in the research will be randomly divided into 4 groups, one group will receive a standard 8 SMT (Stress Management Training) psychological interviews, one group will receive 8 (SMT) psychological interviews and subjects will use an APP together with a CA (Conversational Agent), one group will receive only the APP and the CA, one group will be placed in waiting-list.
  After the closing of the pathway (T2) the subjects will receive the same questionnaires they received at the beginning and again after 3 months (T3).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SMT Group (Active Comparator): This group will receive a standard 8 SMT (Stress Management Training) psychological interviews
  Interventions: Behavioral: SMT
- SMT+CA (Experimental): This group will receive a standard 8 SMT (Stress Management Training) psychological interviews and subjects will use an APP together a CA (Conversational Agent) an Artificial Intelligence.
  Interventions: Behavioral: SMT; Device: App CA
- Only CA (Experimental): This group will receive only an APP together a CA (Conversational Agent) an Artificial Intelligence.
  Interventions: Device: App CA
- Waiting-List (No Intervention): This group will not receive any intervention

INTERVENTIONS:
Behavioral: SMT — Standard 8 SMT (Stress Management Training) psychological interviews.
  Arms: SMT Group; SMT+CA
Device: App CA — An APP together a CA (Conversational Agent).
  Arms: Only CA; SMT+CA

SUMMARY:
The purpose of this study is to identify effective methodologies to help people improve their ability to adapt to psychological stress.

DETAILED DESCRIPTION:
The subjects involved will follow a Stress Management Training (SMT) to learn some techniques to manage stress in the workplace and to increase the effectiveness of the intervention will use an APP and a Conversational Agent (CA) an Artificial Intelligence (AI).

The purpose of the smartphone Application (APP) and CA will be to help people identify their thoughts, help them understand their emotions and the events that generated them.

The data collected and analyzed will be integrated into artificial intelligence to improve understanding of what people are writing.

Based on these analyses, it will be possible to identify the many different variables that interact in cases where a subject shows signs of stress related to adapting to change in the work environment and possible resilience factors that contribute to decreasing the state of stress.

Tests will be administered at the beginning, at the end of the meetings, and 3 months after the end of the sessions. Subjects will be divided into various groups to understand whether APP and CA have a significant impact in increasing psychological well-being and stress coping strategies.

ELIGIBILITY:
Inclusion Criteria:

* whitecollar
* Normal or moderate levels of anxiety and stress
* A sufficient level of education to understand study procedures and be able to communicate with site personnel
* at least 40 to 70 years old

Exclusion Criteria:

* High levels of depression combined with other psychological risk indices (such as suicidal thoughts)
* Current use of narcotics or other substances

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
An improvement of the scales contained in the OSI questionnaire | Up to day 60
  The Occupational Stress Indicator (OSI) test is a validated tool to detect sources of stress, coping styles, and the effects of stress on the job.
An average improvement in Perceived Stress Scale (PSS) test scores | Up to day 60
  The Perceived Stress Scale (PSS) test is a validated test for detecting general stress levels.

SECONDARY OUTCOMES:
An improvement in levels of general psychological well-being Symptom Check List-90-Revised (SCL-90-R) | Up to day 60
  The Symptom Check List-90-Revised (SCL-90-R) test is a validated test for the detection of some psychological scales such as anxiety, depression and the level of general psychological well-being.
An improvement in levels of GAD-7 test scores | Up to day 60
  The GAD-7 test is a validated test for the detection of generalized anxiety disorder. GAD-7 total score for the seven items ranges from 0 to 21. Higher scores mean worse outcome.
An improvement in levels of PHQ-8 test scores | Up to day 60
  The PHQ-8 test is a validated test for the detection of depression. The PHQ-8 is scored just like the PHQ-9 and its total score ranges from 0 to 24. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Ciulli, Principal Investigator — Idego srl
Locations (1):
- Idego srl, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Clinical data obtained from psychological testing and socio-demographic data and any feedback collected during the trial will be shared.
Supporting Information: Study Protocol
Time Frame: Data will be available starting from March 2022 for five years.
Access Criteria: The data available on the research website (www.co-adapt.it). A specific page will be create where researchers can download the raw data to perform any analysis.
URL: https://www.co-adapt.it/research/

REFERENCES:
- [Derived] Danieli M, Ciulli T, Mousavi SM, Silvestri G, Barbato S, Di Natale L, Riccardi G. Assessing the Impact of Conversational Artificial Intelligence in the Treatment of Stress and Anxiety in Aging Adults: Randomized Controlled Trial. JMIR Ment Health. 2022 Sep 23;9(9):e38067. doi: 10.2196/38067. PMID 36149730